CLINICAL TRIAL: NCT01298843
Title: Pharmacokinetics of a Single Dose of Ceftaroline Fosamil in Children Ages Birth to Younger Than 12 Years With Suspected or Confirmed Infection
Brief Title: Study of Blood Levels of Ceftaroline Fosamil in Children Who Are Receiving Antibiotic Therapy in the Hospital
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: P903-21
Record Dates: First submitted 2011-02-15; First posted 2011-02-18 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Infections
Keywords: Confirmed or Suspected Infections
MeSH Terms: conditions — Infections | interventions — Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study of Blood Levels of Ceftaroline Fosamil (Other): Study of Blood Levels of Ceftaroline Fosamil in Children Who Are Receiving Antibiotic Therapy in the Hospital
  Interventions: Drug: Ceftaroline fosamil

INTERVENTIONS:
Drug: Ceftaroline fosamil — Single dose of 15 mg/kg (up to 600 mg) by intravenous infusion

SUMMARY:
The purpose of this study is to assess blood levels of Ceftaroline fosamil in children.

DETAILED DESCRIPTION:
To characterize single dose pharmacokinetics of Ceftaroline fosamil in children.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following inclusion criteria:

* Male or female children with ages from birth to younger than 12 years
* Hospitalized and receiving systemic antibiotic therapy for treatment of a suspected or confirmed infection
* Sufficient intravascular access
* Negative urine pregnancy test
* Written informed consent from parent(s)and verbal informed assent from subject

Exclusion Criteria:

Subjects must NOT meet any of the following exclusion criteria:

* History of any hypersensitivity or allergic reaction to any β-lactam antimicrobial
* Past or current history of epilepsy or seizure disorder
* Moderate or severe renal impairment
* If female, currently pregnant or nursing
* Aspartate aminotransferase, alanine aminotransferase, or total bilirubin level > 3 times upper limit of normal
* Any condition that would make the subject, in the opinion of the Investigator, unsuitable for the study
* Use of probenecid within 3 days prior to dosing
* Receipt of a blood transfusion during the 24-hour period before enrollment

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of Ceftaroline fosamil, plasma concentrations time profile of ceftaroline fosamil by patient, age cohort and dosage level, and Safety and tolerability of ceftaroline fosamil following a single dose of ceftaroline. | Up to 5 days
  This study has 3 primary outcome measures: plasma concentration of ceftaroline fosamil and its metabolites from blood samples after a single dose; PK profile of ceftaroline, and safety, where number of subjects with serious and non-serious adverse events and type of frequency of adverse events will be reported.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Investigational Site, Phoenix, Arizona
  - Investigational Site, Little Rock, Arkansas
  - Investigational Site, Orange, California
  - Investigational Site, San Diego, California
  - Investigational Site, Indianapolis, Indiana
  - Investigational Site, Louisville, Kentucky
  - Investigational Site, Shreveport, Louisiana
  - Investigational Site, Jackson, Mississippi
  - Investigational Site, Omaha, Nebraska
  - Investigational Site, Akron, Ohio
  - Investigational Site, Cleveland, Ohio
  - Investigational site, Toledo, Ohio
  - Investigational Site, Forth Worth, Texas
  - Investigational Site, Morgantown, West Virginia